CLINICAL TRIAL: NCT04180722
Title: A Virtual Transition Intervention for Children and Adults Transitioning to Home Ventilation in Ontario: A Pragmatic Randomized Controlled Trial
Brief Title: Transition to LIVE (Long-term In Home Ventilation Engagement) Study
Acronym: TTLive
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: West Park Healthcare Centre (Other); The Ottawa Hospital (Other); Sunnybrook Health Sciences Centre (Other); London Health Sciences Centre (Other); Children's Hospital of Eastern Ontario (Other); McMaster Children's Hospital (Other); Kingston Health Sciences Centre (Other); Aetonix Systems (Unknown)
Responsible Party: Principal Investigator, Reshma Amin, Staff Physician, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1000000000
Record Dates: First submitted 2019-11-21; First posted 2019-11-27 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Long-term Ventilation at Home
Keywords: Home mechanical ventilation; Ventilator assisted individuals; Virtual Intervention

STUDY DESIGN:
Intervention Model Description: Multicenter, prospective 12 months, 7-centre, pragmatic, parallel group, randomized controlled trial with 1:1 allocation of individuals (children and adults) newly transitioning to Home Mechanical Ventilation (HMV) in Ontario that compares a virtual transition intervention to usual care provided by specialist HMV programs.
Who Masked: Outcomes Assessor
Masking Description: The research coordinator that is consenting the patient and doing the intervention allocation will be different than the research coordinator assessing the outcomes. The outcomes assessor will remain blinded as to whether the participant has received the intervention or not
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants will receive multi-component Virtual Transition Intervention facilitated through the aTouchAway™ platform including the usual care provided by specialist HMV programs.
  Interventions: Device: aTouchAway™ platform
- Control (No Intervention): Usual care will be delivered in accordance with the Canadian Thoracic Society (CTS) clinical practice guidelines and includes scheduled face-to-face clinic visits with the ventilator team with the ventilator team within the first month of starting HMV and then every 3, 6, or 12 months depending on medical stability with additional telephone calls/email contact for equipment trouble shooting and management of intercurrent illnesses as needed.

INTERVENTIONS:
Device: aTouchAway™ platform — Participants will receive multi-component Virtual Transition Intervention. The four components of the intervention comprise: (1) routine virtual clinic visits scheduled at the same frequency as usual care; (2) virtual care plan and action plan for respiratory infection/deterioration and management of ventilator issues; (3) remote, weekly and monthly monitoring of ventilator and cough assist metrics, VAI symptoms, and oxygen saturations; and (4) as needed clinical consultations triggered by identification of abnormal parameters or requested by the VAI or family caregiver.
  Arms: Intervention

SUMMARY:
The rising prevalence of ventilator assisted individuals (VAIs) who depend on Home Mechanical Ventilation (HMV) is an escalating public health challenge with important social and economic implications. VAIs are high cost users of the healthcare system, requiring competent healthcare and family caregivers for successful transition to HMV. The TTLive Study will evaluate the effect of a virtual transition intervention delivered through a virtual care platform, compared to usual care on emergent healthcare utilization, caregiver burden, health cost-effectiveness including cost of family caregiver time, and efficiency of clinical encounters for individuals newly transitioning to HMV.

DETAILED DESCRIPTION:
Ventilator Assisted Individuals (VAIs) on HMVs are an ideal population for a virtual care platform that offers a comprehensive bundle of virtual care solutions, sophisticated enough for the complex care demands of this population. A first complex care demand is the challenging clinical follow ups that impose significant financial and medical costs associated with travel to healthcare appointments, and which can predispose these patients to adverse events during travel periods due to an inability to maintain access to some vital technology such as suctioning.

A second complex care demand is the multiple transitions in care as some VAIs on HMVs move between and within healthcare sectors due to changing health status or care needs, and multi-morbidity. Formalized handovers between providers are lacking. This results in information gaps and additional and sometimes unnecessary time spent by healthcare providers searching for care plan documentation.

A third demand is the lack of timely access to respiratory health professionals experienced in HMV and availability of home follow-up, particularly in the early stages of transition which impedes the transition process.

Virtual Care can be defined as any interaction between patients and/or members of their circle of care, occurring remotely, using any form of communication or information technology, with the aim of facilitating or maximizing the effectiveness and quality of patient care. It includes electronic messaging, tele-consultations and tele-monitoring. The advantages of virtual care include the following: 1) enabling the preconditions for truly empowered patients and patient/family-centered care; 2) overcoming the silos of care, and 3) reducing redundancy within the healthcare system by greater knowledge sharing across healthcare sectors. Virtual care provides an opportunity to make healthcare better by overcoming constraints of distance, cost, and time.

In TTLive Study, a multi-component platform delivered on an electronic tablet developed for complex care management at home is used in partnership with the patient, family and healthcare team to enable the following: 1) virtual home visits; 2) customizable care plans; 3) basic clinical workflows that incorporate reminders, completion of symptom profiles and tele-monitoring, and 4) secure communication via messaging, audio, and video calls. Investigators hypothesize that this virtual transition intervention will reduce emergent healthcare utilization, improve the experience of care, reduce caregiver burden, become more cost-effective than usual care, and enable more efficient use of healthcare provider time.

ELIGIBILITY:
Participant Eligibility Criteria

Inclusion Criteria:

i. Individuals newly initiated (in-hospital or as an outpatient) on a ventilator for HMV prescribed by a participating ventilation program in the previous two months.

ii. Reads, writes and understands English if does not have a caregiver than can do so.

iii. Provides informed consent.

Exclusion criteria:

i. Projected life expectancy of ≤ 2 months. ii. Significant cognitive impairment and absence/inability of a family caregiver to use aTouchAway™ or complete questionnaires.

iii. Uncontrolled psychiatric illness. iv. No internet access (SIM cards and data costs will be covered by the project budget).

v. Currently enrolled in a research study to evaluate another eHealth platform or care coordination.

vi. Plans to move outside of Ontario within the next 12 months.

Caregivers Eligibility Criteria

Caregiver Inclusion Criteria:

i. Primary caregiver of an individual newly initiated (in-hospital or outpatient) on a ventilator for HMV prescribed by a participating clinic in the previous two months; ii. Reads, writes and understands English; and iii. Provides informed consent.

Eligibility Criteria for the Qualitative Interviews

Investigators will exclude those participants:

i. Unable to communicate verbally for the duration of an interview

Inclusion Criteria for Healthcare Providers in the Circle of Care for the Intervention Group

Healthcare provider of an individual from a participating centre i. Use of the aTouchAway for at least five participant encounters ii. Provides informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 444 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2026-01-30 (Actual); Study Completion 2026-01-30 (Actual)

PRIMARY OUTCOMES:
ED Visits: ED visit rates at 12 months determined using health administrative databases | 12 months± 4 weeks
  Using health administrative databases and the Ambulatory Health Care Record-modified
To measure caregiver reported sense of mastery (Pearlin Mastery Scale; scores range up to 28, higher scores = higher mastery), if no caregiver available then patient reported sense of mastery will be utilized | 12 months± 4 weeks
  To measure caregiver reported sense of mastery, an outcome that is often linked to patient empowerment using the Pearlin Self-Mastery Scale, if no caregiver available then patient reported sense of mastery will be utilized

SECONDARY OUTCOMES:
Number of hospital admissions and days in hospital over 6 months using health administrative databases. | 6 months± 4 weeks
  Using health administrative databases and the Ambulatory Health Care Record-modified
Number of hospital admissions and days in hospital over 12 months using health administrative databases. | 12 months ± 4 weeks
  Using health administrative databases and the Ambulatory Health Care Record-modified
Hospital free survival using health administrative data at 6 months. | 6 months ± 4 weeks
  Using health administrative databases and the Ambulatory Health Care Record-modified
Hospital free survival using health administrative data at 12 months. | 12 Months ± 4 weeks
  Using health administrative databases and the Ambulatory Health Care Record-modified
Time to first ED visit and first hospital admission. | 12 months ± 4 weeks
  Using health administrative databases and the Ambulatory Health Care Record-modified
Overall survival at 6 months. | 6 months ± 4 weeks
  Using health administrative databases and the Ambulatory Health Care Record-modified
Overall survival at 12 months. | 12 months ± 4 weeks
  Using health administrative databases and the Ambulatory Health Care Record-modified
Respiratory and non-respiratory causes of death at 6 months. | 6 months ± 4 weeks
  Using health administrative databases and the Ambulatory Health Care Record-modified
Respiratory and non-respiratory causes of death at 12 months. | 12 months ± 4 weeks
  Using health administrative databases and the Ambulatory Health Care Record-modified
Number and type of outpatient specialist visits at 6 months. | 6 months ± 4 weeks
  Using health administrative databases and the Ambulatory Health Care Record-modified
Number and type of outpatient specialist visits at 12 months. | 12 months ± 4 weeks
  Using health administrative databases and the Ambulatory Health Care Record-modified
Number of family physician visits at 6 months. | 6 months ± 4 weeks
  Using health administrative databases and the Ambulatory Health Care Record-modified
Number of family physician visits at 12 months. | 12 months ± 4 weeks
  Using health administrative databases and the Ambulatory Health Care Record-modified
Homecare service use at 6 months. | 6 months ± 4 weeks
  Using health administrative databases and the Ambulatory Health Care Record-modified
Homecare service use at 12 months. | 12 months ± 4 weeks
  Using health administrative databases and the Ambulatory Health Care Record-modified
Change in Zarit Burden Interview Score from baseline to 6 months.The 22 items are assessed on a 5-point Likert scale, ranging from 0 = 'never' to 4 = 'nearly always'. | 6 months ± 4 weeks
  Caregiver Outcome
Change in Zarit Burden Interview Score from baseline to 12 months.The 22 items are assessed on a 5-point Likert scale, ranging from 0 = 'never' to 4 = 'nearly always'. | 12 months ± 4 weeks
  Caregiver Outcome
Change in study participant health related quality of life using the EQ-5D (adults) and ED-5DY (children) change from baseline and 6 months | 6 months ± 4 weeks
  Health Related Quality of Life Outcome
Change in study participant health related quality of life using the EQ-5D (adults) and ED-5DY (children) change from baseline and 12 months | 12 months ± 4 weeks
  Health Related Quality of Life Outcome
Quality of care coordination using Family Experiences with Care Coordination (FECC) for qualitative interview participants only | 6 months ± 4 weeks
  Care Coordination Outcome
Incremental Cost Effectiveness Ratios (ICER) of Virtual Transition intervention compared to usual care in improving patient utility from a societal perspective and using a one-year time horizon | 12 months ± 4 weeks
  Economic Outcome
Mean monthly healthcare costs (public, private and caregiver lost time) over 6 months | 6 months ± 4 weeks
  Economic Outcome: Using health administrative databases and the Ambulatory Health Care Record-modified
Mean monthly healthcare costs (public, private and caregiver lost time) over 12 months | 12 months ± 4 weeks
  Economic Outcome: Using health administrative databases and the Ambulatory Health Care Record-modified
Encounter time spent by clinicians over 12 months measured using the Care Coordination Measurement Tool | 12 months ± 4 weeks
  HealthCare Provider Outcome
Process Measure Outcomes | 12 months ± 4 weeks
  n(%) of 5 clinic visits conducted virtually as opposed to face to face
Process Measure Outcomes | 12 months ± 4 weeks
  n (%) of virtual data downloads available for the virtual clinic visits
Process Measure Outcomes | 12 months ± 4 weeks
  n(%) participants that completed the virtual care plan within 6 weeks after intervention initiation
Process Measure Outcomes | 12 months ± 4 weeks
  n (%) of the 52 weekly check-ins completed
Process Measure Outcomes | 12 months ± 4 weeks
  n(%) of the 12 monthly S3-NIV check-ins completed
Process Measure Outcomes | 12 months ± 4 weeks
  number of ad hoc questions/concerns in which healthcare team contacted via the platform
Process Measure Outcomes | 12 months ± 4 weeks
  number of status yellow monitoring alerts initiated based on the weekly and monthly symptom monitoring and time to alert being addressed by a member of the circle of care
Process Measure Outcome- Qualitative Interviews | 6 months ± 4 weeks
  Qualitative interviews to explore the experience with the aTouchAway intervention by study participants, caregivers and healthcare providers
Process Measure Outcome- Site focus Groups | 24 months ± 4 weeks
  Our LIVE study data has shown reduction in ED visits due to the pandemic and since ED Visits are the primary outcome for TtLIVE, as a process measure, we will conduct a one-time focus group to generate a hierarchy of important study primary and secondary outcomes with participating sites.
  Site focus groups: Every participating site will get an opportunity to participate in a 30-60-minute focus group to discuss and rank outcomes relevant to their practice over zoom

CONTACTS AND LOCATIONS:
Overall Officials: Reshma Amin, MD, MSc, Principal Investigator — The Hospital for Sick Children; Louise Rose, PhD, Principal Investigator — King's College London; Andrea Gershon, MD, MSc, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (8):
- Canada (8):
  - McMaster Children's Hospital, Hamilton, Ontario
  - Children's Hospital, London Health Sciences, London, Ontario
  - London Health Sciences Center, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - Sunnybrook Health Sciences Center, Toronto, Ontario
  - West Park Healthcare Centre, York, Ontario

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Amin R, Gershon A, Buchanan F, Pizzuti R, Qazi A, Patel N, Pinto R, Moretti ME, Ambreen M; TtLIVE Group; Rose L. The Transitions to Long-term In Home Ventilator Engagement Study (Transitions to LIVE): study protocol for a pragmatic randomized controlled trial. Trials. 2022 Feb 7;23(1):125. doi: 10.1186/s13063-022-06035-z. PMID 35130935